CLINICAL TRIAL: NCT05594017
Title: Behavioral and Pharmacological Manipulation of Time Cell Activity in the Human Mesial Temporal Lobe
Brief Title: Pharmacological Modulation of Brain Oscillations in Memory Processing
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Bradley Lega, ASSOC PROFESSOR - Neurological Surgery, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STU 022018-005; R01NS125250 (NIH)
Record Dates: First submitted 2022-10-17; First posted 2022-10-26 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Epilepsy; Seizures; Cognitive Impairment, Mild; Memory Disorders; Memory Loss
Keywords: oscillatory changes; cholinergic antagonist; muscarinic antagonist
MeSH Terms: conditions — Epilepsy; Seizures; Cognitive Dysfunction; Memory Disorders | interventions — Scopolamine

STUDY DESIGN:
Intervention Model Description: Patients are randomized to scopolamine or saline solution by the pharmacy upon drug receipt. Both researchers and patients are blinded to which session receives pharmaceutical versus placebo administration. Each of the patients receive scopolamine or placebo on Day 1 and Day 2 before completing tasks at critical time points to parse encoding and retrieval.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Scopolamine (0.4mg) (Experimental): Subjects will receive a dose of scopolamine (0.4mg) on each day. Approximately 15 minutes after administration, the participant will then complete either an episodic or a spatial memory task session.
  If the patient completed the sham session already, this session will take place the day following the initial session, or at least four half-lives after the first session.
  Interventions: Drug: Scopolamine (0.4mg)
- Placebo (Placebo Comparator): Subjects will receive saline (0.4mg) via IV on each day. Approximately 15 minutes after administration, the participant will then complete either an episodic or a spatial memory task session.
  If the patient completed the scopolamine session already, this session will take place the day following the initial session, or at least four half-lives after the first session.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Scopolamine (0.4mg) — Patient receives a dose of scopolamine (0.4mg) via IV fifteen minutes prior to spatial or episodic memory task/completion.
  Arms: Scopolamine (0.4mg)
Drug: Placebo — Patient receives a dose of saline via IV fifteen minutes prior to spatial or episodic memory task/completion.
  Arms: Placebo

SUMMARY:
The goal of this study is to learn about the effects of scopolamine (an anticholinergic drug) on areas of the brain involved in memory, and changes it may have on brain activity. The investigators will do this by testing epileptic patients who are already undergoing intracranial surgery for seizure monitoring, and measuring the activity from the brain areas being assessed.

The main questions it aims to answer are 1) whether scopolamine changes memory activity solely at encoding (the time when the person perceives and determines to remember an item or event) as has previously been found, or if it also can selectively impact retrieval (when the item or event which has been processed is recalled or remembered), and 2) what the nature of the brain activity changes is.

Participants will complete two treatment arms. One of these will be with the drug, and the other will be with a saline solution, so that the participants are unaware which session the actual drug has been received. Patients will complete a verbal and/or spatial task each of the two days. An anesthesiologist will administer either the drug or the saline at a critical point which addresses both of the research questions.

Researchers will compare the brain activity between the two treatment arms to determine what brain activity changes, and at what time point during memory formation.

DETAILED DESCRIPTION:
Patient Identification : The study team plans to recruit adult patients who are undergoing invasive electroencephalographic (EEG) monitoring as part of a standard clinical procedure for the treatment of pharmacologically resistant epilepsy at UT Southwestern. Patients are identified from the pool of patients presented at the epilepsy management conference and approached when presented to the clinic for evaluation for seizure surgery.

Study Procedures: Participation takes place only during the time that the electrodes are surgically in place. Active participation will end when the electrodes are removed. The subject may decline to participate in cognitive testing sessions at any given time during intracranial monitoring hospitalization and are informed of the right to leave the study at any time. The neuropsychological tasks described below will be administered by key personnel on the study. The data will be de-identified and converted to signal data for processing and analysis. Study personnel, excluding the PI (aka 'experimenters') will perform analysis.

Once patients are in the epilepsy monitoring unit (EMU), subjects will be randomized to receive either a dose of scopolamine (0.4mg) or saline (sham) via IV. Approximately 15 minutes after administration, the participant will then complete either an episodic or a spatial memory task session. The following day, or at least four half-lives after the first session, the participant will receive the alternative agent not given the first day. For example, if the patient received Scopolamine the first day, then the saline (sham) is received the second day, and vice versa. The participants will then complete an additional episodic or spatial memory task session approximately 15 minutes after administration. ,

Day 1: Randomized to receive either Scopolamine or saline (sham); Complete episodic or spatial memory task session Day 2: Receives alternate agent from day 1; Completes episodic or spatial memory task session

The time delay between sessions will stay consistent whether scopolamine or saline was administered during the first session. Participants will not be administered more than one dosage during a single session.

The attending physician and nurse will know whether scopolamine or saline are being administered, but the participant will not know if what is being administered until after both sessions are completed.

The participant's attending nurse will administer intravenous scopolamine and/or saline.

The effects of scopolamine will make true patient blinding difficult, but for this, the study will be modeled on fMRI tasks in which administration was blinded.

Physiologic Monitoring: Patients in the epilepsy monitoring undergo EKG and pulse oxygen monitoring at all times as part of routine care and this will not be interrupted during the study period. A board-certified anesthesiologist will be present during the beginning of the period to treat any cardiopulmonary complications using standard techniques, if necessary, and will be immediately available within the hospital to respond with any other concerns.

Overview of Memory Testing : The cognitive experiments typically last 30-75 minutes and are without physical risk to participants. Depending on patient enthusiasm, multiple trials can be performed with intervening rest breaks, and sessions may last several hours. Participants may stop and resume anytime. Participants, who are generally hospitalized for 1-2 weeks because of epilepsy, choose how frequently to take part in the experimental sessions. By participating in cognitive tasks, patients incur no additional medical or surgical risk, and in fact often report that the game-like testing protocols provide relief from the boredom of awaiting seizures. Within each session, the participants are allowed to take frequent breaks to avoid fatigue. Testing can and will be immediately interrupted for any health-care-related needs.

Episodic (Free Recall) or Spatial Memory Task: The study team's existing paradigm has used Free Recall for testing episodic memory. In this task, participants study lists of items and attempt to recall as many words as possible from each list. Lists are comprised of words or nameable pictures. A computer controls stimulus presentation and records participants' responses. Following the last item of each list, participants are either asked to recall the list immediately, or are first given a series of simple arithmetic problems to solve (this end-of-list distracter task serves to reduce the large advantage accorded to end-of-list items during recall). There are approximately 10-12 words or items in one list. Participants are then given a period of between 30 seconds and three minutes to recall list items in any order. The participants' responses are digitally recorded by the computer and anonymously stored for later analysis. In order to address additional questions of interest with regards to oscillations in the hippocampal areas, and how these react to real and imagined navigation, the study team is adding a spatial memory task, in which participants will be requested to navigate in a virtual environment from one location to another, then simulate the same navigation in the mind visually. For each actual navigation, the simulation process is repeated. Logs are made of the time spent visualizing, as well as several catch trials where subjects move the controller to mimic the actual navigation. These are then correlated with the EEG files. The inclusion of both tasks allows the study team to address both novel questions regarding the oscillations in the hippocampus in navigation sequences, as well as allowing further data collection on this existing protocol.

Collection of iEEG data: All EEG data are collected for clinical purposes by clinicians, using a computerized EEG collection system. In this study, the study team will copy these data, strip the data of any confidential information, and analyze the raw traces of EEG. Synchronization of the experimental computer with the iEEG signals is accomplished by sending an optically isolated pulse to an input on the EEG recording system. The testing computer will send a stereotyped train of pulses (five or ten 10-millisecond (ms) pulses separated by 10 ms) at the start and end of each experimental block plus a single 10-ms pulse at regular intervals of one second. This train of pulses enables the iEEG record to synchronize itself with the testing computer. The starting train will make it easy to locate the beginning of an experimental session. In this way, the two clocks are resynchronized frequently, preventing event times from drifting significantly throughout the course of an experiment.

ELIGIBILITY:
Patient inclusion criteria:

1. Age 18 - 55 years, all races/ethnicities, and both genders are eligible.
2. Candidates for pre-operative evaluation using stereo intracranial electrodes and admission to the Epilepsy Monitoring Unit (EMU) as determined independently by the patient's treating physician as part of the patient's routine medical care.
3. Able to read, understand, and provide written, dated informed consent prior to screening.
4. In good general health, aside from a history of epilepsy, as ascertained by medical history, physical examination (PE), clinical laboratory evaluations, and ECG.
5. Body mass index between 18-35 kg/m2.

Patient exclusion criteria:

1. Has a clinically significant abnormality on the screening physical examination that might affect safety, study participation, or confound interpretation of study results according to the study physician.
2. Female that is pregnant, breastfeeding, or has a positive pregnancy test at screening or baseline. Note that pregnant patients are excluded from undergoing iEEG generally and all patients undergo a positive screening urine test for drugs of abuse at screening: cannabinoids, cocaine, amphetamines, barbiturates, opiates not otherwise explained by their prescribed medications.
3. History of renal insufficiency.
4. Unstable cardiac syndrome or active cardiac symptoms.
5. Patients with liver failure.
6. Patients with BPH.
7. Patients with autoimmune neuropathy.
8. Patients with uncontrolled hyperthyroidism.
9. Patients with a history of dementia.
10. Patient with a history of delirium after using transdermal scopolamine.
11. History of narrow-angle glaucoma.
12. History of pyloric obstruction or paralytic ileus.
13. History of myasthenia gravis, obstructive uropathy, porphyria, or myasthenia gravis.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Memory-related changes in brain electrical activity in participants from baseline at Day 1 post-intervention (approx. within 1-3 hrs) | Baseline, at Day 1 post-intervention (approx. within 1-3 hrs)
  Memory-related changes in brain electrical activity in participants from baseline at post-intervention (approx. within 1-3 hrs) is measured by comparing the Free recall memory tasks with the electrical readings collected across all bandwidths, but focusing on primarily theta changes.
Memory-related changes in brain electrical activity in participants from baseline at Day 2 post-intervention (approx. within 1-3 hrs) | Baseline, at Day 2 post-intervention (approx. within 1-3 hrs)
  Memory-related changes in brain electrical activity in participants from baseline at post-intervention (approx. within 1-3 hrs) is measured by comparing the Free recall memory tasks with the electrical readings collected across all bandwidths, but focusing on primarily theta changes.
Memory-related changes in brain electrical activity in participants from baseline at Day 1 post-intervention (approx. within 1-3 hrs) | Baseline, at Day 1 post-intervention (approx. within 1-3 hrs)
  Memory-related changes in brain electrical activity in participants from baseline at post-intervention (approx. within 1-3 hrs) is measured by comparing the Spatial memory tasks with the electrical readings collected across all bandwidths, but focusing on primarily theta changes.
Memory-related changes in brain electrical activity in participants from baseline at Day 2 post-intervention (approx. within 1-3 hrs) | Baseline, at Day 2 post-intervention (approx. within 1-3 hrs)
  Memory-related changes in brain electrical activity in participants from baseline at post-intervention (approx. within 1-3 hrs) is measured by comparing the Spatial memory tasks with the electrical readings collected across all bandwidths, but focusing on primarily theta changes.
Memory-related changes in brain electrical activity in participants from baseline at Day 1 post-intervention (approx. within 1-3 hrs) | Baseline, at Day 1 post-intervention (approx. within 1-3 hrs)
  Memory-related changes in brain electrical activity in participants from baseline at post-intervention (approx. within 1-3 hrs) is measured by comparing the serial recall memory tasks with the electrical readings collected across all bandwidths, but focusing on primarily theta changes.
Memory-related changes in brain electrical activity in participants from baseline at Day 2 post-intervention (approx. within 1-3 hrs) | Baseline, at Day 2 post-intervention (approx. within 1-3 hrs)
  Memory-related changes in brain electrical activity in participants from baseline at post-intervention (approx. within 1-3 hrs) is measured by comparing the serial recall memory tasks with the electrical readings collected across all bandwidths, but focusing on primarily theta changes.
Memory-related changes in brain electrical activity in participants from baseline at Day 1 post-intervention (approx. within 1-3 hrs) | Baseline, at Day 1 post-intervention (approx. within 1-3 hrs)
  Memory-related changes in brain electrical activity in participants from baseline at post-intervention (approx. within 1-3 hrs) is measured by comparing the associative recognition memory tasks with the electrical readings collected across all bandwidths, but focusing on primarily theta changes.
Memory-related changes in brain electrical activity in participants from baseline at Day 2 post-intervention (approx. within 1-3 hrs) | Baseline, at Day 2 post-intervention (approx. within 1-3 hrs)
  Memory-related changes in brain electrical activity in participants from baseline at post-intervention (approx. within 1-3 hrs) is measured by comparing the associative recognition memory tasks with the electrical readings collected across all bandwidths, but focusing on primarily theta changes.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley C Lega, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No